CLINICAL TRIAL: NCT00205712
Title: Prevention of NMDA Antagonist-induced Psychosis and Memory Impairment in Children
Brief Title: Prevention of N-methyl-D-aspartate (NMDA) Antagonist-induced Psychosis in Kids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NARSAD - Kids; 01-0886 (Other: Washington University IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Psychoses, Substance-Induced
Keywords: NMDA antagonist-induced psychosis; Children; Memory Impairment; Decreased cognitive function; Increased memory impairment
MeSH Terms: conditions — Psychoses, Substance-Induced; Memory Disorders | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine plue saline (Placebo Comparator): Ketamine without dexmedetomidine
  Interventions: Drug: Ketamine
- Ketamine plus dexmedetomidine (Experimental): Ketamine infusion plus dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine — Ketamine without dexmedetomidine
  Other Names: Ketanest; Ketaset; Ketalar
  Arms: Ketamine plue saline
Drug: Dexmedetomidine — Ketamine plus dexmedetomidine
  Other Names: Precedex
  Arms: Ketamine plus dexmedetomidine

SUMMARY:
Ketamine, an FDA approved anesthetic agent, is becoming the sedative/analgesic of choice for emergency sedation in children because it causes deep sedation with minimal respiratory depression in comparison to other available agents. However, emergence reactions are an important adverse effect of ketamine, characterized by transient changes in cognitive function, dissociation and mild schizophrenia-like symptoms. These cognitive and behavioral effects are dose-dependently induced by ketamine and other antagonists of the N-methyl-D-aspartate (NMDA) glutamate receptor. NMDA receptor hypofunction can disinhibit excitatory (cholinergic/glutamatergic) projections in key areas of the brain, and this has been proposed to explain key features of schizophrenia. Several treatments that block excessive excitatory transmitter release have also been shown to prevent cognitive and behavioral effects of ketamine-induced NMDA receptor hypofunction in humans. Alpha-2 adrenergic agonists, which can presynaptically inhibit acetylcholine release, can prevent mild ketamine-induced behavioral and cognitive symptoms in healthy human adults. However, this prevention strategy has not been evaluated in children. Children currently receive clinically-indicated treatment with the NMDA antagonist, ketamine, and this age group is an important target for pharmacological strategies aimed at the prevention of schizophrenia. This application proposes a double-blind, placebo-controlled, randomized trial to test the safety and effectiveness of dexmedetomidine, an FDA approved alpha-2 adrenergic agonist, in preventing ketamine-induced mental symptoms in children. Planned primary analyses will evaluate effects of the hypothesized prevention treatment on clinical and cognitive variables using analysis of variance (ANOVA). The proposed experiments are relevant to future prevention trials for individuals at risk for schizophrenia, and to preventing adverse effects of NMDA antagonist anesthetic agents (ketamine, nitrous oxide).

DETAILED DESCRIPTION:
The proposed study will be conducted using existing dedicated clinical and research space in St. Louis Children's Hospital's Emergency Department, Pediatric Clinical Research Center (PCRC), and Orthopedic Clinic. This project has 3 major aims and 1 exploratory aim addressed by a prospective randomized blinded placebo controlled drug trial to test whether a pharmacological strategy can prevent NMDA receptor hypofunction-induced behavioral and cognitive dysfunction in pre- and post-pubertal children. Based on previous preclinical and clinical research on the effects and blockade of the effects of ketamine and similar compounds, the study investigators have carefully selected a dose of the alpha-2 adrenergic agonist dexmedetomidine that will permit this study to be conducted with low risk to enrolled subjects who are undergoing clinically-indicated ketamine sedation for forearm fracture reduction.

General Experimental Design: This project will test the safety and effectiveness of dexmedetomidine for preventing ketamine-induced behavioral and cognitive symptoms in healthy human children undergoing clinically indicated ketamine sedation for forearm fracture reduction.

Aims 1 and 2 will be addressed by randomized, blinded administration of dexmedetomidine or saline placebo to ketamine-sedated subjects to test the efficacy of dexmedetomidine in preventing ketamine-induced behavioral and cognitive changes during recovery from sedation.

Aim 3 will be addressed by comparing between the subjects randomized to receive dexmedetomidine or saline placebo measurements of distress and frequency of adverse cardiopulmonary effects during sedation, fracture-reduction, and recovery.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to St. Louis Children's Hospital's Emergency Department who require reduction of an acute forearm fracture will be recruited for enrollment if they satisfy the following:

1. Age 7-17 years, inclusive;
2. Are psychiatrically healthy (i.e. have never been under the care of a psychiatrist or taken psychiatrically active medications);
3. Meet American Society of Anesthesiologist (ASA) Class I and II criteria (I=healthy, II=chronic disease under good control);
4. Have had no prior fracture reduction or ketamine administration;
5. Present for care when research assistants are present (Monday-Friday, 09:00-23:00); and
6. Have a home telephone or ready means of establishing telephone contact.

All subjects and their parent/guardian will give Washington University Human Studies Committee approved written informed assent and consent prior to participation.

Exclusion Criteria:

1. Solid food intake 2 hours or less before procedure;
2. Compromised cardiorespiratory function; central nervous system, hepatic, or renal abnormality;
3. History of psychosis in patient or first degree relative;
4. Currently taking medications that stimulate or depress mental function, e.g. methylphenidate for attention deficit hyperactivity disorder or drugs of abuse;
5. History of allergy or adverse reaction to alpha-2 adrenoreceptor agonist drugs, e.g. clonidine.

These exclusion criteria relate to contraindications for use of the agents employed in the study. Criteria 1, 2, 3 and 4 are current routine practice for ketamine sedations.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2003-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Newcomer, M.D., Principal Investigator — Washington University School of Medicine and Florida Atlantic University
Locations (1):
- Washington University School of Medicine, Psychiatry Dept., St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Alone: Ketamine without dexmedetomidine
Period: Overall Study
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.2) | 10.9 (2.4) | 11 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Ratings Scale (BPRS) Positive Symptom Subscale Score
Description: Participant received behavioral ratings before medication and during medication for the primary analysis comparison. This is an observer-scale with a value range from 0-6 (0=no symptoms 6=worst symptoms)
Time Frame: Before Ketamine, During Ketamine
Population: Completers analysis per protocol. Two participants were missing some data at either the before ketamine or during ketamine time point.
Measure: Mean (Standard Deviation); unit: Scale of 0-6
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine
Number analyzed (Participants) | 20 | 18
Scale of 0-6
  BPRS Positive symptom subscale-before medication | 0.00 (0.00) | 0.00 (0.00)
  BPRS Positive symptom subscale-during medication | 1.40 (2.37) | 1.00 (1.41)

2. Secondary Outcome: Visual Analog Scale (VAS) Pain Intensity
Description: Pain intensity was measured on a scale of 1-10 (1=lowest pain intensity, 10=highest pain intensity) in participants before medication, during medication, post medication and 1 week follow up.
Time Frame: Before Ketamine, During Ketamine, Post Ketamine and 1 Week Follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scale of 1-10
Groups:
- Ketamine Plus Dexmedetomidine: Ketamine infusion with dexmedetomidine
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine
Number analyzed (Participants) | 18 | 18
Scale of 1-10
  VAS Pain-Before Medication | 4.72 (1.93) | 4.03 (2.38)
  VAS Pain-Before Cognitive Testing | 2.75 (1.65) | 2.89 (1.78)
  VAS Pain-After Cognitive Testing | 2.61 (1.33) | 4.08 (1.85)
  VAS Pain-1 Week F/U | 1.33 (0.59) | 1.76 (1.64)

3. Secondary Outcome: Visual Analog Scale (VAS) Anxiety Rating
Description: Anxiety was measured on a scale of 1-10 (1=lowest pain intensity, 10=highest pain intensity) in participants before medication, during medication, post medication and 1 week follow up.
Time Frame: Before Ketamine, During Ketamine, Post Ketamine, 1 week follow up
Measure: Mean (Standard Deviation); unit: Scale of 1-10
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine
Number analyzed (Participants) | 20 | 18
Scale of 1-10
  VAS Anxiety-Before Medication | 5.0 (2.43) | 5.0 (2.35)
  VAS Anxiety-Before Cogntive Testing | 1.67 (0.97) | 2.53 (1.58)
  VAS Anxiety-After Cognitive Testing | 1.71 (1.14) | 3.00 (2.04)
  VAS Anxiety-1 Week Follow Up | 1.56 (1.20) | 2.06 (1.82)

ADVERSE EVENTS:
Arm/Group | Ketamine Alone | Ketamine Plus Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Alone (N=20) | Ketamine Plus Dexmedetomidine (N=20)
Sedation (Nervous system disorders) | 19 (19) | 19 (19)
Nausea/Vomiting (Gastrointestinal disorders) | 5 (5) | 12 (12)
headache (Nervous system disorders) | 3 (3) | 7 (7)
Dizziness (Nervous system disorders) | 11 (11) | 11 (11)
Difficulty Walking (Nervous system disorders) | 4 (4) | 4 (4)
Trouble Breathing (General disorders) | 2 (2) | 1 (1)
Visual Hallucinations (Nervous system disorders) | 6 (6) | 6 (6)
Unpleasant Dreams (Nervous system disorders) | 4 (4) | 2 (2)
Numbness (Nervous system disorders) | 15 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No